CLINICAL TRIAL: NCT00466687
Title: A Phase II Trial of Tarceva (Erlotinib) and Avastin (Bevacizumab) in the Treatment of Patients With Metastatic Melanoma
Brief Title: Erlotinib and Bevacizumab in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey A. Sosman, MD, Professor of Medicine; Director, Melanoma and Tumor Immunotherapy, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC MEL 0418; VU-VICC-MEL-0418; VU-IRB-040468
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Melanoma
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Erlotinib Hydrochloride; In Situ Hybridization, Fluorescence; Gene Expression Profiling; Immunologic Techniques; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental): Tarceva and Avastin:
  * Tarceva: 150mg PO, days 1-28
  * Avastin: 10mg/kg, IV infusion, days 1,15 Regimen will be repeated every 28 days = 1 course
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride; Genetic: fluorescence in situ hybridization; Genetic: gene expression analysis; Other: immunologic technique; Other: laboratory biomarker analysis; Procedure: biopsy

INTERVENTIONS:
Biological: bevacizumab — 10mg/kg, slow IV infusion, Days 1 and 14
  Other Names: Avastin
Drug: erlotinib hydrochloride — 150mg PO qd
  Other Names: Tarceva
Genetic: fluorescence in situ hybridization — Targeting multiple genetic aberrations in isolated tumor cells.
Genetic: gene expression analysis — gene expression analysis
Other: immunologic technique — immunologic technique
Other: laboratory biomarker analysis — laboratory biomarker analysis
Procedure: biopsy — biopsy

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving erlotinib together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving erlotinib together with bevacizumab works in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate, response duration, and frequency of progression-free survival at 6 months in patients with stage IV melanoma treated with erlotinib hydrochloride and bevacizumab.
* Determine objective responses in patients treated with this regimen.

Secondary

* Determine the overall safety and tolerability of this regimen in these patients.
* Evaluate tissue blocks for EGFR by monoclonal antibody H11 (DAKO) or fluorescence in situ hybridization(FISH)7p12-specific probe-overexpression or amplification in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib hydrochloride once daily on days 1-28 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tissue collection to analyze EGFR by monoclonal antibody H11 (DAKO) or fluorescence in situ hybridization (FISH) 7p12-specific probe-overexpression or amplification. Biological markers AKT, MAPK, p27, p21, CD13, CD34, and factor VIII are also measured.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Measurable Stage IV melanoma
* Easter Cooperative Oncology Group (ECOG) Performance Status must be 0-1
* Good organ function as demonstrated by, Creatinine <2.mg/dl, AST or ALT <5 times upper limit of normal for subjects with documented liver metastases; <2.5 times the upper limit of normal (ULN) for subjects without evidence of liver metastases, bilirubin<2.0mg/dl,, absolute neutrophil count (ANC)>1500/ul, platelets>75k/ul, hemoglobin (Hgb)>9 (may be transfused to obtain)
* Prior therapy: adjuvant interferon (IFN) allowed; no more than one prior regimen for advanced stage IV disease
* Patients must have a life expectancy of >3 months
* Patients with brain metastases are eligible only if they fulfill the following: resected or stereotactic treatment a minimum of 3 months previously and no active CNS disease since then; brain metastases treated greater than 6 months ago without evidence of progression or hemorrhage, <1cm in size per lesion (up to 3 lesions), and off all steroids
* Patients may not have received other agents, either investigational or marketed, which act by either EGFr inhibition or anti-angiogenesis mechanisms. Other epidermal growth factor receptor (EGFR) inhibitors include (but are not limited to): Iressa, erbitux, CI-1033. Angiogenesis inhibitors include (but are not limited to): SU5416, SU6668, SU 0122348, CP547632, VEGF Trap, anti-integrin αVβ3.
* Recovered from toxicity of major surgery (4 wks), chemotherapy or biologic therapy (4 wks), and/or radiation therapy (2 wks)
* No active other malignancy within 12 months
* No active systemic infection
* Over age of 18 years and signed IRB approved informed consent

Exclusion Criteria:

* Subjects meeting any of the following criteria (3.2.2-3.2.16) are ineligible for study entry
* Compromised renal or hepatic function as defined by Creatinine >2.0mg/dl, aspartate transaminase (AST) or alanine transaminase (ALT) >5 times upper limit of normal for subjects with documented liver metastases; >2.5 times the upper limit of normal (ULN) for subjects without evidence of liver metastases
* Patient may not be part of any other investigational studies
* internationalized normal ratio (INR) > 1.5
* Patients with PEG or G-tube are ineligible.
* Major surgical procedure, open biopsy; or significant traumatic injury within 28 days, or anticipation of need for major surgical procedure during the course of the study
* Any non-healing wound, ulcer, or bone fracture.
* Any clinical evidence or history of a bleeding diathesis or coagulopathy.
* Patients with a history of deep vein thrombosis or thromboembolic disease within the past 6 months.
* History of acute myocardial infarction within 6 months. In addition, patients are ineligible if they have clinically significant cardiovascular disease ((e.g., uncontrolled hypertension [blood pressure of >160/110 mmHg on medication], New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac dysrhythmia requiring medication, or peripheral vascular disease (Grade II or greater)
* Patients with > 1+ proteinuria will have 24-hour urine collection; for protein. Patients with ≥ 1gm protein/24 hrs will be excluded
* If child bearing age must not be pregnant or nursing and use methods to prevent pregnancy
* History or evidence upon physical examination of central nervous system (CNS) disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, or history of stroke)
* Inability to comply with study and/or follow-up procedures
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-09; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Sosman, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study remained open from 09/15/2004 to 1/27/2006.
Pre-assignment Details: 36 patients consented to be in the study, two were determined not eligible.
Groups:
- Therapeutic Intervention: Patients receive pemetrexed disodium IV and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for up to 4 courses. If patient progresses before receiving 4 courses of treatment, treatment will be discontinued and patient will proceed to surgery.
Period: Overall Study
Arm/Group | Therapeutic Intervention
Started | 34
Completed | 0
Not Completed | 34
Not completed — Adverse Event | 1
Not completed — Other complicating illness | 3
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression | 29

BASELINE CHARACTERISTICS:
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response
Description: Per Response Evaluation Criteria in Solid Tumor (RECIST): Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: At 6 months
Population: Patients for whom a response could be determined. Three patients were not available for measurement of response: no data (2) and toxicity (1).
Measure: Number; unit: participants
Groups:
- Tarceva/Avastin: Study drugs are administered on a 28-day cycle for 6 cycles: Tarceva 150 mg by mouth per day and Avastin 10 mg/kg of body weight intravenously (IV) on days 1 and 15.
Arm/Group | Tarceva/Avastin
Number analyzed (Participants) | 31
participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 14
  Progressive Disease | 15

2. Secondary Outcome: Time to Disease Progression.
Description: Time from on study date to date of progression in months, if the progression happened in the patient. Disease progression is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions with reference to the smallest sum LD since treatment began or the appearance of one or more new lesions.
Time Frame: up to one year after off-study date
Population: Patients with disease progression. Six patients were not available for determination to progression: no data (5) and toxicity (1).
Measure: Median (Full Range); unit: Months
Arm/Group | Tarceva/Avastin
Number analyzed (Participants) | 28
Months | 3 [1 to 12]

3. Secondary Outcome: Progression-free Survival at 6 Months
Description: Patients with Progression-free survival at 6 months
Time Frame: 6 months
Population: Those patients who were progression-free at 6 months from study entry. No date of progression was available for 7 patients
Measure: Number; unit: participants
Groups:
- Therapeutic Intervention: Study drugs are administered on a 28-day cycle: Tarceva 150 mg by mouth per day and Avastin 10 mg/kg of body weight intravenously (IV) on days 1 and 15.
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 27
participants | 7 [1 to 28]

4. Secondary Outcome: Number of Patients With Each Worst-grade Toxicity Response
Description: Number of patients with worst-grade toxicity at each of five grades following National Cancer Institute Common Toxicity Criteria with grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening/disabling, 5 = death.
Time Frame: Day 1 of each 28-day cycle for 6 cycles (168 days)
Population: Patients who received the study drug and who experienced a toxicity. Eleven patients did not experience any toxicity and are therefore not included in the analyzed population for this outcome measure.
Measure: Number; unit: participants
Groups:
- Tarceva/Avastin: Study drugs are administered on a 28-day cycle: Tarceva 150 mg by mouth per day and Avastin 10 mg/kg of body weight intravenously (IV) on days 1 and 15.
Arm/Group | Tarceva/Avastin
Number analyzed (Participants) | 23
participants
  No. of patients with worst-grade toxicity of 1 | 3
  No. of patients with worst-grade toxicity of 2 | 12
  No. of patients with worst-grade toxicity of 3 | 7
  No. of patients with worst-grade toxicity of 4 | 1
  No. of patients with worst-grade toxicity of 5 | 0

ADVERSE EVENTS:
Arm/Group | Therapeutic Intervention
Serious Adverse Events (participants affected / at risk) | 10/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Intervention (N=34)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Pain - tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Edema limb-right leg (Cardiac disorders) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 2 (2)
apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
confusion (Renal and urinary disorders) | 1 (1)
death not associated with CTCAE term-disease progression NOS (General disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (3)
fatigue (General disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
muscle weakness (not due to neuropathy) extra-occular (Eye disorders) | 1 (1)
muscle weakness (not due to neuropathy) unable to walk (Musculoskeletal and connective tissue disorders) | 1 (1)
muscle weakness (not due to neuropathy) whole body (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (5)
pain abdomen (Gastrointestinal disorders) | 2 (3)
pain back (Musculoskeletal and connective tissue disorders) | 1 (2)
pain buttock, pelvis (Musculoskeletal and connective tissue disorders) | 1 (1)
pain extremity, limb (Musculoskeletal and connective tissue disorders) | 1 (1)
pain neck (Musculoskeletal and connective tissue disorders) | 1 (2)
colon perforation (Gastrointestinal disorders) | 1 (1)
pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
platelets (Blood and lymphatic system disorders) | 1 (1)
pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
somnolence (Nervous system disorders) | 1 (1)
sweating (Skin and subcutaneous tissue disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Intervention (N=34)
alkaline phosphatase (Investigations) | 5 (16)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (20)
ALT, SGPT (Investigations) | 3 (5)
anorexia (Metabolism and nutrition disorders) | 13 (51)
AST, SGOT (Investigations) | 4 (10)
bilirubinemia-imcreased (Hepatobiliary disorders) | 2 (2)
Cardiac general-other (Cardiac disorders) | 3 (9)
cholesterol, serum-high (Investigations) | 2 (2)
constipation (Gastrointestinal disorders) | 5 (18)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (32)
diarrhea (Gastrointestinal disorders) | 10 (64)
fatigue (General disorders) | 18 (104)
Fever (in the absence of neutropenia, with neutropenia defined as ANC < 1.0 x 10e9/L (General disorders) | 2 (8)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 4 (22)
glucose, serum-high (Metabolism and nutrition disorders) | 9 (24)
heartburn, dyspepsia (Gastrointestinal disorders) | 4 (19)
hemoglobin (Investigations) | 6 (22)
hemorrhage, pulmonary/upper respiratory-lung (Respiratory, thoracic and mediastinal disorders) | 2 (8)
hypertension (Vascular disorders) | 6 (41)
infection with unknown-bladder (urinary) (Infections and infestations) | 2 (21)
insomnia (Psychiatric disorders) | 3 (19)
magnesium, serum low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 (11)
mood alteration-anxiety (Psychiatric disorders) | 2 (4)
mood alteration-depression (Psychiatric disorders) | 4 (20)
mucositis/stomatitis-oral cavity (Infections and infestations) | 2 (2)
musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 2 (9)
nausea (Gastrointestinal disorders) | 8 (55)
pain-abdomen NOS (Gastrointestinal disorders) | 3 (9)
pain-back (Musculoskeletal and connective tissue disorders) | 2 (6)
pain-extremity. limb (Musculoskeletal and connective tissue disorders) | 3 (6)
pain-head/headache (Nervous system disorders) | 4 (14)
pain-other (General disorders) | 3 (12)
pain-tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6)
potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (6)
proteinuria (Renal and urinary disorders) | 3 (36)
pruritis (Skin and subcutaneous tissue disorders) | 5 (57)
rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (22)
rash acne/acneiform (Skin and subcutaneous tissue disorders) | 12 (91)
renal/genitourinary-other (Renal and urinary disorders) | 2 (12)
sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (7)
sweating/diphoresis (Skin and subcutaneous tissue disorders) | 2 (9)
voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3 (21)
vomiting (Gastrointestinal disorders) | 4 (12)
weight loss (Metabolism and nutrition disorders) | 3 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes